CLINICAL TRIAL: NCT05640596
Title: Antenatal Corticosteroid Therapy: Which Impact on Birth Parameters?
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENARD Emeline, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2021PI166
Record Dates: First submitted 2022-07-12; First posted 2022-12-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Growth Retardation
Keywords: Antenatal corticosteroid therapy; newborn; growth
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- exposed group (121 patients): Extrated from the population of full-term newborns (> 36 weeks of amenorrhea + 6 days) between 2014 and 2020 at the Regional Maternity Hospital of Nancy who received at least one course of betamethasone before 34 weeks of amenorrhea for a threat of preterm delivery.
  Exposure to an antenatal corticosteroid therapy was defined as the administration of at least one course of betamethasone (i.e. two doses of 12 mg, 24 hours apart). in intramuscular, before 34 weeks of amenorrhea, for a threat of premature delivery.
  Interventions: Drug: Betamethasone
- nonexposed group (242 patients): came from the population of full-term newborns (> 36 weeks of amenorrhea + 6 days) between 2014 and 2020 at the Regional Maternity Hospital of Nancy who who had not been exposed to antenatal steroid therapy. Two controls were selected for a case, appaired on the month and year of birth and on the sex of the case patient.

INTERVENTIONS:
Drug: Betamethasone
  Groups: exposed group (121 patients)

SUMMARY:
Use of antenatal corticosteroids therapy has increased since the 2000s. The benefits of such a therapy on premature newborns are scientifically and internationally recognized.

Nevertheless, few studies have been conducted to investigate the impact of this antenatal corticosteroid therapy on full-term newborns (> 36 weeks' gestation).

The aim of this study is to compare the birth parameters of full-term newborns exposed or not to antenatal corticosteroid therapy.

DETAILED DESCRIPTION:
All children included in the study were born at the Regional Maternity Hospital of Nancy between January 1, 2014 and December 31, 2020.

One hundred and twenty-one of them were exposed during pregnancy to antenatal corticosteroids therapy and constitute the exposed arm, whereas 242 were not and constitute the non-exposed arm.

Data were collected retrospectively regarding history of pregnancy, birth parameters and neonatal adaptation.

ELIGIBILITY:
Inclusion Criteria:

* all children exposed to an antenatal corticosteroid therapy before 34 weeks of amenorrhea because of a threat of premature delivery
* only full-term newborns

Exclusion Criteria:

* all children exposed to an antenatal corticosteroid therapy before 34 weeks of amenorrhea for other reasons

Max Age: 12 Months | Sex: All
Age Groups: Child
Study Population: All children included in the study were born at the Regional Maternity Hospital of Nancy between January 1, 2014 and December 31, 2020.
  One hundred and twenty-one of them were exposed during pregnancy to antenatal corticosteroids therapy and constitute the exposed arm, whereas 242 were not and constitute the non-exposed arm.
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of an antenatal corticosteroid therapy on head growth. | Birth
  head circumference

SECONDARY OUTCOMES:
Evaluate the impact of an antenatal corticosteroid therapy on fetal weight | Birth
  birth weight
Evaluate the impact of an antenatal corticosteroid therapy on fetal growth | birth
  birth lenght
Evaluate the impact of an antenatal corticosteroid therapy on neonatal adaptation : APGAR score for each patient | birth
  APGAR score
Evaluate the impact of an antenatal corticosteroid therapy on risk of hypoglycemia : number of patients with neonatal hypoglycémia | first 5 days
  hypoglycemia
Evaluate the impact of an antenatal corticosteroid therapy on risk of hypocalcemia : number of patients with hypoglycemia | first 5 days
  hypocalcemia
Evaluate the impact of an antenatal corticosteroid therapy on neonatal outcome : number of days of hospitalisation after birth | first 5 days
  day of hospitalisations after birth
Evaluate the impact of an antenatal corticosteroid therapy on eating disorders (number of patients with difficulty to drink) | first 5 days
  eating disorders

REFERENCES:
- [Derived] Best C, Hascoet JM, Jeanbert E, Morel O, Baumann C, Renard E. Impact of corticosteroid exposure on preterm labor in neonates eventually born at term. J Perinatol. 2024 Feb;44(2):195-202. doi: 10.1038/s41372-023-01831-0. Epub 2023 Dec 1. PMID 38040875